CLINICAL TRIAL: NCT06274138
Title: The Enchanting Symphony of Haptonomy's Impact on Attachment and Spousal Harmony for Women Conceiving Through Infertility Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HAPTONOMY
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-07

CONDITIONS: Infertility
Keywords: haptonomy; pregnancy; attachment; marital adjustment; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- haptonomy (Experimental): Pregnant women in the intervention group will complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. Information will be given that Haptonomy will consist of five sessions. Haptonomy will be applied by the researcher together with the partner. Each session will last for 40 minutes. The effectiveness and continuity of sessions will be planned between 3 to 7 days. One week after completing the five sessions of haptonomy, pregnant women will again complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. The completion of the scales will take approximately 10-15 minutes.
  Interventions: Behavioral: haptonomy
- control (No Intervention): Explanation of the purpose of the study will be provided to pregnant women and their partners, obtaining verbal and written consent. Pregnant women in the control group will complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. The completion of the scales will take approximately 10-15 minutes.

INTERVENTIONS:
Behavioral: haptonomy — Pregnant women in the intervention group will complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. Information will be given that Haptonomy will consist of five sessions. Haptonomy will be applied by the researcher together with the partner. Each session will last for 40 minutes. The effectiveness and continuity of sessions will be planned between 3 to 7 days. One week after completing the five sessions of haptonomy, pregnant women will again complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. The completion of the scales will take approximately 10-15 minutes.
  Arms: haptonomy

SUMMARY:
Pregnancies resulting from infertility treatment are considered normal and 'low-risk' in some countries, they often entail significant stress. Prenatal attachment may be experienced differently by parents conceiving through fertility interventions. The rising prevalence of fertility treatments is associated with increased risks such as preterm birth, low birth weight, and perinatal mortality for pregnancies achieved through infertility treatments. Beyond medical implications, post-infertility treatment pregnancies can induce high levels of anxiety and a perception of pregnancy as risky, affecting individuals psychologically. The transition to parenthood after infertility treatment can be psychologically challenging.

Healthy prenatal attachment in expectant mothers fosters the development of a healthy role as both mother and father. Maternal bonding is closely tied to a woman's mental health during the prenatal period and her commitment to her baby. Similarly, prenatal bonding with the father sheds light on the emotional connection developing between the father and the unborn child. Active participation in prenatal experiences, such as attending ultrasound appointments or discussing parenting plans, contributes to a stronger sense of attachment for fathers and establishes a positive foundation for future bonding. Supportive partner relationships during pregnancy enhance paternal bonding and emphasize the importance of a collaborative approach to prenatal care for both parents. The prenatal period is critical for fathers to establish an early emotional connection with their unborn children, laying a positive groundwork for postnatal bonding.

Various interventions aim to enhance communication between parents and augment prenatal attachment. One such practice is haptonomy-haptotherapy. Haptotherapy focuses on restoring emotional connections, especially with one's own body. It helps individuals recognize their emotional capacities and allows them to experience these capacities through insightful conversations, therapeutic touch, and skill exercises. In the context of pregnancy, haptonomy involves physical contact between the pregnant woman, her partner, and the unborn baby. Advocates of haptonomy believe that this touch-based communication can strengthen the bond between parents and the baby, promote a sense of security, and positively influence the pregnancy experience.

Haptonomy is thought to contribute positively to the psychological well-being of women during pregnancy, birth, and the postpartum period, potentially preventing mental health issues and enhancing the health of both mother and baby. It is emphasized that haptonomy is a distinct practice focused on enhancing communication between parents and the baby. Existing literature suggests that haptonomy can increase emotional bonding during the prenatal period and may be effective for parents showing low attachment. Studies indicate that touch communication develops from the second month, involving vibrations for communicating with the fetus, ultimately increasing bonding through haptonomy. Furthermore, haptonomy is reported to enhance both spousal and parental attachment, as demonstrated in a study emphasizing increased attachment for fathers with their partners and children.

Despite documented benefits of haptonomy in various patient groups, from cancer patients undergoing chemotherapy to pregnant women and those with chronic pain, limited research exists on haptotherapy for pregnant women. This study aims to investigate the impact of partner-administered haptonomy on prenatal attachment and marital adjustment in pregnant women. Conducted through a randomized controlled experimental design, the study seeks to provide evidence by enhancing prenatal attachments in both mothers and fathers.

Research Hypotheses:

H0-1: The application of haptonomy by partners has an effect on maternal attachment in pregnant women.

H1-1: The application of haptonomy by partners does not have an effect on maternal attachment in pregnant women.

H0-2: The application of haptonomy by partners has no effect on paternal attachment in pregnant women.

H1-2: The application of haptonomy by partners has an effect on paternal attachment in pregnant women.

H0-3: The application of haptonomy by partners has no effect on marital adjustment in pregnant women.

H1-3: The application of haptonomy by partners has an effect on marital adjustment in pregnant women.

DETAILED DESCRIPTION:
Study Design A randomly clinical trial with pre-session and post-session, was conducted. Participants and blindly and randomly allocated to the intervention group (haptonomy) or the control group, using a random number generator by the researcher.

Participants and procedures The population of the study consists of pregnant women and their partners who are being followed up at the Başkent University Ankara Hospital IVF Center between December 25, 2023, and December 25, 2024, and have become pregnant through infertility treatment, ranging from the 20th to the 28th week of pregnancy. The sample of the study will consist of pregnant women who meet the inclusion criteria and agree to participate in the research. The sample size was calculated by conducting a power analysis using the G*Power program and referring to previous studies. According to the power analysis, with an effect size of 0.70 and a 5% margin of error, a minimum sample size of 68 individuals (34 experimental, 34 control) is required to achieve a power of 0.80. Considering possible data losses, a total of 76 individuals (38 experimental, 38 control) will be included in the study. The randomization of the sample will be determined by entering the total number of cases into the program at the URL address https://www.randomizer.org. Before entering the data into the program, it is assumed that set 1 will represent the control group, and set 2 will represent the intervention group. The program will determine the random order of the cases comprising the sample group through the randomization method. Participants eligible for this study must have successfully achieved pregnancy through infertility treatment. They should currently be in the 20th to 28th week of pregnancy and must be living together with their spouse. Those who fall outside the 20th to 28th week of pregnancy, individuals living separately from their spouse, and those experiencing a high-risk pregnancy will not be included in the study.

Outcome measures Sociodemographic form Sociodemographic form, which was constructed by the researcher based on the literature, included questions about the week of pregnancy, age, education, socioeconomic status, and questions to assess fetal-parent communication.

Marital Adjustment Scale (MAS):

The MAS, developed by Locke and Wallace (1959) and adapted to Turkish by Tutarel-Kışlak (1999), consists of 15 items. Scores on the scale increase from discordance to harmony. The lowest adjustment score is 1, and the highest is 60. The scale assesses happiness levels in marriage, with questions 2 and 9 measuring disagreements between spouses based on specified criteria.

Prenatal Attachment Inventory (PAI):

Developed in 1993 by Muller and Mercer, the PAI aims to understand pregnant women's thoughts and feelings throughout pregnancy and determine their attachment levels to the baby during the prenatal period. The Turkish version's reliability is established by Yılmaz and Beji (2013). The scale consists of items scored on a 1-4 Likert scale.

Antenatal Father Attachment Scale (AFAS):

The AFAS, developed by John Condon (1993), comprises 16 items as a 5-point Likert scale to measure fathers' emotions, thoughts, attitudes, and behaviors related to their unborn babies. The Turkish validity and reliability study is conducted by Benli and Aksoy Derya (2019).

Study Variables:

The study will measure the mean scores of the prenatal attachment scale for pregnant women. Mean scores of the antenatal father attachment scale will be assessed for fathers. The marital adjustment scale will be utilized to determine the mean scores for both mothers and fathers. The independent variable in this study is the application of Haptonomy.

Data Collection procedure:

The study will involve pregnant women and their partners receiving haptonomy in the intervention group and those in the control group continuing routine follow-ups. Comparison of attachment and marital adjustment scores between the intervention and control groups will be conducted. Both groups will undergo the following procedures:

Intervention Group:

Explanation of the purpose of the study and information about Haptonomy will be provided to pregnant women and their partners, obtaining verbal and written consent. Pregnant women in the intervention group will complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. Information will be given that Haptonomy will consist of five sessions. Haptonomy will be applied by the researcher together with the partner. Each session will last for 40 minutes. The effectiveness and continuity of sessions will be planned between 3 to 7 days. One week after completing the five sessions of haptonomy, pregnant women will again complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. The completion of the scales will take approximately 10-15 minutes.

Control Group:

Explanation of the purpose of the study will be provided to pregnant women and their partners, obtaining verbal and written consent. Pregnant women in the control group will complete the Prenatal Attachment Scale and Marital Adjustment Scale, and fathers will complete the Antenatal Father Attachment Scale and Marital Adjustment Scale through face-to-face interviews. The completion of the scales will take approximately 10-15 minutes.

Statistical Analysis:

Data will be analyzed using the licensed IBM SPSS 23 software. Descriptive statistics such as numbers, percentages, means, and standard deviations will be used. Normal distribution will be assessed using the Kolmogorov-Smirnov test. For binary group comparisons, the independent samples t-test or Mann-Whitney U Analysis will be used based on normality. For within-group comparisons, the paired samples t-test or Wilcoxon analysis will be applied for normal and non-normal distributions, respectively. Results will be evaluated at a 95% confidence interval, and significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy after infertility treatment
* 28-36 weeks of gestation
* Living with his/her spouse

Exclusion Criteria:

* Outside the 28-36th gestational week
* Living separately from his/her spouse
* Having a risky pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Marital adjustment score | pre-intervention, two weeks after the intervention, four weeks after the intervention
  Marital Adjustment Scale will be used to assess this outcome measure. Scores in the scale increase from incompatibility to compatibility. The lowest compliance score is 1 and the highest score is 60.
Prenatal attachment score | pre-intervention, two weeks after the intervention, four weeks after the intervention
  Prenatal Attachment Inventory will be used to assess this outcome measure. A minimum of 21 and a maximum of 84 points can be obtained from the scale. As the scale score increases, attachment level increases.
Father attachment score | pre-intervention, two weeks after the intervention, four weeks after the intervention
  Antenatal Father Attachment Scale will be used to assess this outcome measure. A minimum of 16 and a maximum of 80 points are obtained from the scale. As the scale score increases, attachment level increases.

CONTACTS AND LOCATIONS:
Overall Officials: İlçim Ercan Koyuncu, Study Director — Baskent University; Cansu Akdağ Topal, Study Director — Baskent University
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No